CLINICAL TRIAL: NCT02193256
Title: Pilot Trial of Varenicline and Prazosin to Treat Heavy Drinking Smokers
Brief Title: Varenicline + Prazosin for Heavy Drinking Smokers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1402013410; K05AA014715 (NIH)
Record Dates: First submitted 2014-07-14; First posted 2014-07-17 (Estimated); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Cigarette Smoking; Alcohol Use Disorders
Keywords: varenicline; prazosin; cigarette smoking; alcohol drinking; sleep; dreams
MeSH Terms: conditions — Cigarette Smoking; Alcoholism; Alcohol Drinking | interventions — Varenicline; Prazosin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Varenicline plus Prazosin (Active Comparator): Varenicline: .5mg for 3 days then 1mg daily for 4 days (Week 1) then 2mg daily thereafter (Weeks 2-3). Prazosin: 1mg for 3 days, then 3mg for 4 days (Week 1), (2) 6mg for 3 days, then 8mg for 4 days (Week 2), and (3) 8mg (Week 3).
  Interventions: Drug: Varenicline; Drug: Prazosin
- Varenicline plus Placebo (Placebo Comparator): Varenicline: .5mg for 3 days then 1mg daily for 4 days (Week 1) then 2mg daily thereafter (Weeks 2-3). Placebo: placebo will be given instead of prazosin (Weeks 1-3)
  Interventions: Drug: Varenicline; Drug: Placebo

INTERVENTIONS:
Drug: Varenicline — Titrated over 1 week to a maximum dose of 2mg/day
  Other Names: Chantix
Drug: Prazosin — Titrated over 3 weeks to a maximum dose of 8mg/day
  Other Names: Minipress
  Arms: Varenicline plus Prazosin
Drug: Placebo
  Arms: Varenicline plus Placebo

SUMMARY:
The purpose of this study is to examine the effect of varenicline and prazosin on smoking, drinking, and sleep among cigarette smokers who report heavy alcohol use. Varenicline is an FDA approved smoking cessation medication. Some smokers report sleep problems when taking varenicline. This study will test whether using prazosin, which is an FDA-approved blood pressure medication, in combination with varenicline reduces sleep problems that can be associated with using varenicline for smoking cessation. In addition, the study will examine the combined effects of these medications on smoking and drinking.

Hypothesis: Varenicline plus prazosin will result in lower rates of vivid dreams and insomnia symptoms/sleep discontinuity than varenicline alone prior to the 3-day practice quit attempt.

Hypothesis: Varenicline plus prazosin will result in lower rates of vivid dreams and insomnia symptoms/sleep discontinuity than varenicline alone during the 3-day practice quit attempt.

DETAILED DESCRIPTION:
The study comprises an 8-week double-blind, within-subjects, crossover design of varenicline (up to 2mg per day) plus either prazosin (up to 8mg per day) (V+P) or placebo (V) with 20 heavy drinking smokers. Each medication phase is 3 weeks with a 2-week medication washout in between. Participants are asked to make a practice quit attempt for 3 days the last week of each medication phase.

This is an exploratory study to look at two primary aims:

1. Evaluate the effect of prazosin on sleep disturbance caused by varenicline in heavy drinking smokers prior to quitting smoking.

   Hypothesis: V+P will result in lower rates of vivid dreams and insomnia symptoms/sleep discontinuity than V alone.
2. Evaluate the effect of prazosin on sleep disturbance caused by varenicline during smoking cessation in heavy drinking smokers.

Hypothesis: V+P will result in lower rates of vivid dreams and insomnia symptoms/sleep discontinuity than V alone We will also investigate the combined effects of prazosin and varenicline on smoking behavior (i.e., smoking urge) and alcohol consumption (i.e., drinks per drinking day) as exploratory aims.

ELIGIBILITY:
Inclusion Criteria:

1. at least 18 years of age;
2. current smoker [quantity of ≥ cigarettes per smoking day, frequency of ≥3 times per week, and urinary cotinine ≥2 on NicAlert dipstick;
3. at least 4 occasions of heavy drinking in the past 30 days [5 or 4 standard drinks per occasion for males and females, respectively];
4. no history of severe alcohol withdrawal syndrome;
5. no new onset of psychiatric illness or psychotropic medications in last 90 days;
6. no severe psychiatric illness [schizophrenia, bipolar disorder] or PTSD;
7. no substance dependence other than nicotine, alcohol or marijuana;
8. no medical contraindications for varenicline or prazosin;
9. are willing to take medication and wear portable sleep monitoring devices;
10. no risk for sleep apnea syndrome;
11. able to read and write in English;
12. not interested in quitting smoking immediately.

Exclusion Criteria:

1. unable to complete the informed consent;
2. do not meet criteria for heavy drinking;
3. do not meet criteria for current smokers;
4. unable to read/understand English;
5. exhibit serious psychiatric illness (i.e. schizophrenia, bipolar disorder, severe major depression, panic disorder, borderline personality disorder), organic mood or mental disorders by history of psychological examination;
6. meet criteria for alcohol dependence in past 12 months that is clinically severe;
7. meet criteria for drug dependence in the last 12 months aside from marijuana, nicotine and alcohol;
8. are seeking to quit smoking immediately;
9. report current psychosis or suicidality;
10. are a female of childbearing potential who is pregnant, nursing, or not practicing effective contraception (oral, injectable, or implantable contraceptives, intrauterine device, or barrier method with spermicide);
11. exhibit current, clinically significant physical disease or abnormality based on medical history, physical examination, or routine laboratory evaluation including:

    1. any unexplained elevations in liver enzymes (i.e. transaminases, bilirubin);
    2. clinically significant, unstable cardiovascular disease/uncontrolled hypertension;
    3. hepatic or renal impairment;
    4. severe obstructive pulmonary disease;
    5. diabetes mellitus requiring insulin or certain oral medications (i.e. sulfonylureas) and an A1C hemoglobin test score of >7 for participants not prescribed these medications;
    6. baseline systolic blood pressure higher than 150 mm Hg of diastolic blood pressure higher than 95 mm Hg; (g) are scheduled for cataract surgery; (h) have a diagnosis of narcolepsy;
12. have a history of cancer (except treated basal cell or squamous cell carcinoma of the skin)
13. have a history of clinically significant allergic reactions;
14. have used any psychotropic drug in the past month, except individuals who are on a stable dose of a Selective Serotonin Reuptake Inhibitor for at least two months;
15. intend to donate blood or blood products during the treatment phase of the study;
16. have a Body Mass Index (calculated as weight in kilograms divided by the square of height in meters) less than 15 or greater than 28 or weight less than 45 kg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-07; Primary Completion 2015-01 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Effect of prazosin on sleep disturbance caused by varenicline prior to quitting smoking | Two weeks
  Sleep disturbance will be measured using self-report questionnaires (Insomnia Severity Index, Pittsburgh Sleep Quality Index, Pittsburgh Sleep Diary, Dream Quality Questionnaire) and objective sleep-monitoring devices.
Effect of prazosin on sleep disturbance caused by varenicline during smoking cessation | One week
  Sleep disturbance will be measured using self-report questionnaires (Insomnia Severity Index, Pittsburgh Sleep Quality Index, Pittsburgh Sleep Diary, Dream Quality Questionnaire) and objective sleep-monitoring devices.

OTHER OUTCOMES:
Number of cigarettes smoked | Three weeks
  The investigators will compare the combined effects of prazosin and varenicline on the number of cigarettes smoked with varenicline alone.
Number of drinks per drinking day | Three weeks
  The investigators will compare the combined effects of prazosin and varenicline on alcohol consumption (i.e., number of drinks per drinking day) with varenicline alone as an exploratory aim.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M Fucito, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States